CLINICAL TRIAL: NCT04110496
Title: A Phase 1b Open-Label Single Dose Safety, Tolerability, and Pharmacokinetics Study of RTX-134 in Adults With Phenylketonuria
Brief Title: Safety and Tolerability of RTX-134 in Adults With Phenylketonuria
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was discontinued by the Sponsor
Sponsor: Rubius Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTX-134-01
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RTX-134 (Experimental): Escalating doses of RTX-134 will be administered by intravenous infusion one time
  Interventions: Drug: RTX-134

INTERVENTIONS:
Drug: RTX-134 — RTX-134 is a cellular therapy containing AvPAL

SUMMARY:
This study will evaluate the safety and tolerability of RTX-134 in adult patients with PKU.

DETAILED DESCRIPTION:
This is a Phase 1b first-in-human trial in adult subjects with PKU. The primary objective of this study is to evaluate the safety and tolerability of RTX-134 following intravenous administration of a single dose. RTX-134 consists of allogeneic human red cells expressing the AvPAL (Anabaena variabilis phenylalanine ammonia lyase) gene inside the cell. The trial is designed to determine a preliminary dose and inform a dosing schedule that is deemed safe, tolerable, and potentially effective. Four dose levels are planned, additional dose levels may be explored. Following administration, subjects will be monitored until 28 days after last detection of RTX-134. Detection of RTX-134 will be evaluated using multiple pharmacokinetic (PK) and pharmacodynamic (PD) assessments including measurement of trans-cinnamic acid (tCA).

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older with:

   1. A clinical diagnosis of PKU, and
   2. Average blood phenylalanine level ≥ 600 µmol/L based on 2 assessments up to 3 weeks apart during the 6-month period before Day 0 (per available data)
2. Stable diet, including medical formula
3. Must be a man or a woman not of childbearing potential and agree to use adequate contraception throughout and for one year following study participation.
4. Adequate organ function
5. Negative antibody detection on type and screen and no evidence of clinical hemolysis

Exclusion Criteria

1. Known hypersensitivity to any component of study treatment
2. Prior treatment with Pegaliase
3. Start of sapropterin dihydrochloride within 3 weeks of study dosing
4. Use of an investigational agent within 28 days of study dosing
5. Concurrent participation in an interventional trial involving ongoing treatment, including placebo.
6. Infections requiring antimicrobial treatment within 7 days of study dosing
7. Chronic infections, such as HIV, hepatitis B, or untreated hepatitis C
8. Conditions that may alter survival of red blood cells, (e.g., autoimmune diseases, splenectomy, etc)
9. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of RTX-134 as measured by frequency of treatment emergent adverse events | Baseline to 28 days after last detection of RTX-134
To correlate dose with percent reduction in serum phenylalanine levels relative to baseline | Baseline to 28 days after last detection of RTX-134
To determine a preliminary dose to achieve serum phenylalanine levels < 600 µmol/L | Baseline to 28 days after last detection of RTX-134
To determine a preliminary dose to achieve serum phenylalanine levels < 360 µmol/L | Baseline to 28 days after last detection of RTX-134
To evaluate the pharmacokinetics of RTX-134 as measured by presence of AvPal expressing red cells, AvPAL protein in red cells and serum, and AvPAL enzymatic activity. | Baseline to 28 days after last detection of RTX-134

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No